CLINICAL TRIAL: NCT05971563
Title: Amino Acid Kinetics of GMP-AA Vs. Phenylalanine-free Amino Acids Compared with Natural Protein in Healthy Adults Volunteers
Brief Title: Amino Acid Kinetics of GMP-AA in Healthy Human Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Birmingham Women's and Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 281421
Record Dates: First submitted 2023-07-13; First posted 2023-08-02 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2023-07

CONDITIONS: Phenylketonurias
MeSH Terms: conditions — Phenylketonurias | interventions — Caseins

STUDY DESIGN:
Intervention Model Description: A three-way, randomized, controlled, open-label, crossover, single-dose clinical trial in healthy adult volunteers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Casein (Active Comparator)
  Interventions: Dietary Supplement: Casein
- Glycomacropeptide (Active Comparator)
  Interventions: Dietary Supplement: CGMP-AA
- L- amino acids (Active Comparator)
  Interventions: Dietary Supplement: L-amino acids

INTERVENTIONS:
Dietary Supplement: Casein — Natural protein
  Arms: Casein
Dietary Supplement: L-amino acids — Synthetic amino acids based protein substitute for Phenylketonuria
  Arms: L- amino acids
Dietary Supplement: CGMP-AA — Glycomacropeptide based protein substitute for Phenylketonuria
  Arms: Glycomacropeptide

SUMMARY:
Children with phenylketonuria (PKU) are treated with a special diet supplemented with a synthetic protein based on amino acids. These have a poor taste and are inefficiently used by the body. A different type of synthetic protein, called glycomacropeptide is being tried in PKU. It tastes better than amino acids but it requires the addition of some extra amino acids which may worsen how well it is absorbed compared with traditional amino acid supplements. We will perform a 3-part trial in healthy adult volunteers to compare amino acids vs glycomacropeptide protein with a 'normal protein' (casein) to examine the absorption properties of these proteins. Volunteers will take one dose of each of the protein sources on 3 different days. Blood and urine samples will be collected examining the rate of absorption of amino acids over 5 hours on each study day.

DETAILED DESCRIPTION:
In the USA, casein glycomacropeptide (CGMP), a low phenylalanine (Phe) 64-amino acid peptide derived from cheese whey, is widely promoted as a low Phe protein substitute in phenylketonuria (PKU). Protein substitute is composed of non-essential and essential amino acids which replace natural protein in the diet in order to enable normal growth and suppression of blood Phe levels.

It is suggested that CGMP has a slower absorption than usual protein substitute based on amino acids only (amino acids-AA). This compositional change may enhance protein utilization leading to improved blood Phe control. In PKU, any protein substitute that has its absorption closer to the normal 'physiological state' should be advantageous but pure CGMP is lacking in several essential and conditionally essential amino acids (e.g. tyrosine, leucine, tryptophan, histidine). To ensure that CGMP is safe for PKU, it is supplemented with deficient AA (CGMP-AA). Evidence from 'normal' nutritional research suggests that adding AA to natural protein (similar to CGMP-AA), worsens rather than improves efficiency of protein absorption. It is essential to ascertain if CGMP-AA enhances, worsens or has the same absorption when compared with traditional AA substitutes, particularly when prescribing CGMP-AA for children and maternal PKU. The investigators aim to perform a three-part, randomized, controlled, trial in healthy adult volunteers comparing absorption of CGMP-AA (study product 1) vs. AA (study product 2) vs. normal protein (casein) (study product 3). After overnight fasting, healthy volunteers will consume a standard dose of each of the study products. Over the course of 4 hours, plasma AA will be monitored 8 times and this will provide greater insight into the kinetic absorption of CGMP-AA in PKU. The investigators hope these results will add to existing safety and efficacy data about using CGMP-AA in PKU.

ELIGIBILITY:
Inclusion Criteria:

* Male and female healthy subjects without PKU;
* 18 to 50 years of age;
* Female subjects with a negative urine pregnancy test prior to entry into the study and who are practicing an adequate method of birth control during the study;
* Good general health status proven by medical history and clinical laboratory values within normal limits or considered not clinically significant by the investigator;
* Non-smokers or not current smokers;
* Body mass index (BMI) between 18 and 30 kg/m2 and weight (kg)
* No existence of disorders or any comorbidity.
* Willing to follow the study protocol and to take the study products;
* Able to understand study procedures and sign informed consent.

Exclusion Criteria:

* History of alcohol or drugs abuse;
* Smokers;
* Women who are pregnant, breast feeding, or planning to become pregnant during the course of the study;
* Received an investigational drug or device within 30 days (or 5 half-lives, whichever is longer) of dosing;
* Existence of any disorder, food allergy or comorbidity (clinically significant including gastrointestinal, renal, pulmonary, hepatic, cardiovascular and endocrine disorders) - to be decided by investigator from medical history;
* Current illness or infection that could interfere with the study;
* Use of laxatives;
* Use of antibiotics in the last 3 months;
* Use of medication that could influence protein metabolism (like growth hormone, anabolic steroids, hormone replacement) - to be judged by the investigator;
* Participation in any clinical trial in the last 3 months;
* Blood donation within the past 3 months;
* On a medically prescribed diet;
* Unable to follow the study protocol or provide consent;
* Unable to take or tolerate one of the study products.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Total EAA concentrations | 240 minutes for each protein
  To compare the total EAA concentrations after oral ingestion of one dose of three different protein supplements: cGMP-AA vs. AA only vs. casein.
Mean CMAX | 240 minutes for each protein
  Mean CMAX within 240 minutes of ingestion of each of the 3 proteins
AUC of EAA's | 240 minutes for each protein
  AUC of EAA's within 240 minutes of ingestion of each of the 3 proteins

SECONDARY OUTCOMES:
Curve characteristics (Cmax) | 240 minutes for each protein
  Curve characteristics (Cmax) of the following quantities:
  * LNAA;
  * BCAA;
  * Total AA;
  * Tyrosine;
  * Phenylalanine;
  * Urea;
  * Insulin.
Curve characteristics (AUC) | 240 minutes for each protein
  Curve characteristics (AUC) of the following quantities:
  * LNAA;
  * BCAA;
  * Total AA;
  * Tyrosine;
  * Phenylalanine;
  * Urea;
  * Insulin.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All materials, information (oral or written) and unpublished documentation provided to the Investigators (or any company/institution acting on their behalf), including this protocol and the patient Case Report Forms, are the exclusive property of the Research team and may not be given or disclosed, either in part or in whole, by any person to any third party without the prior express consent of the research team. Potential and recruited patients will be identified by a unique study number with only the local research staff having the corresponding list of full patient identifiers, which should be kept secure. CRFs will be labelled with patient initials and their unique study number. Laboratory results shall be labelled similarly having had patient-identifiable details removed. All unpublished information shall be kept confidential and shall not be published or disclosed to a third party without the prior written consent of the research team.